CLINICAL TRIAL: NCT06251128
Title: Community Stroke Self-management Program for Rural Dwelling African American Stroke Survivors
Brief Title: Community Stroke Self-management Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-09-5982-A
Record Dates: First submitted 2023-11-09; First posted 2024-02-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Blood Pressure
Keywords: Stroke; Community; Aging; Blood pressure; Self management
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single Group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-management (Experimental): This group of participants will be given education and will be taught about overcoming the barriers to a healthy lifestyle and medication adherence. No drugs or devices will be administered to the participants/
  Interventions: Behavioral: Stroke Self management Program

INTERVENTIONS:
Behavioral: Stroke Self management Program — Our educational and behavioral program includes an educational component, problem-solving to overcome barriers to a healthy lifestyle, activities of daily living, and management of medications.
  No drugs or devices will be delivered to the participants
  Other Names: Behavioral

SUMMARY:
This pilot project aims develop a need-based community stroke self-management program that would improve the stroke self-management self-efficacy and competencies among African American stroke survivors living in rural Alabama. This study is a mixed-methods study to collect data related to the needs of these individuals and develop a need-based intervention based on the actual needs/ preferences of our target population. The specific aims are to assess the needs, access barriers, existing resources for a stroke self-management program; and develop a Community Stroke Self-management Program for improving stroke survivors' abilities to manage their medication adherence, diet, Physical Activity (PA) requirements, symptoms, and psychological distress to better meet their needs, expectations, and preferences. Another aim is to examine the feasibility and acceptability of delivering the CSSP after tailoring the proposed intervention in Aim 2a) among the AA chronic stroke survivors living in rural Alabama.

DETAILED DESCRIPTION:
Stroke is a leading cause of mortality and morbidity. African American (AA) populations have a higher prevalence of stroke than whites do. The lack of resources leads to substantial physical, social, and psychological burdens and makes self-management more challenging, hence putting these individuals at high risk for secondary chronic conditions. This is especially prominent among underserved populations including AA living in the black belt of rural Alabama due to the additional factors related to their socio-demographic characteristics. This pilot project aims develop a need-based community stroke self-management program that would improve the stroke self-management self-efficacy and competencies among African American stroke survivors living in rural Alabama. This is a mixed-methods study to collect data related to the needs of these individuals and develop a need-based intervention based on the actual needs/ preferences of the target population. The specific aims are to assess the needs, access barriers, existing resources for a stroke self-management program; and develop a Community Stroke Self-management Program for improving stroke survivors' abilities to manage their medication adherence, diet, Physical Activity (PA) requirements, symptoms, and psychological distress to better meet their needs, expectations, and preferences. The study also aim to examine the feasibility and acceptability of delivering the CSSP after tailoring our proposed intervention in Aim 2a) among the AA chronic stroke survivors living in rural Alabama. Conducting this study would help to have a sustainable intervention with minimal need of healthcare workers for its online delivery, potentially it would have high scalability and a high economic impact in the long run. Therefore, this project is vital for meeting the unique needs of this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* History of Stroke
* High blood pressure condition
* African American
* Age 50 and above

Exclusion Criteria:

-Low cognition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Southampton Score Self Management Questionnaire | 3 months
  Questionnaire;
  Each item on the Southampton Score Self-Management Questionnaire has a minimum score of 1 and a maximum score of 6. A higher score means better Self-management competency following a Stroke.
  The mean of the scores on this questionnaire will be computed for reporting overall scores on this measure.
Hypertension Self-care Activity Level Effects | 3 months:
  Questionnaire; Each item on self-care activity for management of Hypertension has a minimum score of 0 and a maximum score of 7. A higher score means a better Hypertension Self-care Activity Level.
  The mean of the scores on this questionnaire will be computed for reporting overall scores on this measure.
Hypertension Knowledge Level Scale Test | 3 months
  Questionnaire;
  Each item on the Hypertension Knowledge Level Scale has a minimum score of 1 and a maximum score of 5.
  Higher scores on this scale mean a better Hypertension Knowledge Level.
  The mean of the scores on this questionnaire will be computed for reporting overall scores on this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mudasir Andrabi, Ph D, Study Director — The University of Alabama
Locations (1):
- The Hale County extension Office, Greensboro, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified and uploaded to the NIA data sharing repository on a quarterly basis. Data to be shared includes the self-reported data on questionnaires including demographic questionnaire, Stroke self-management competencies questionnaire, data collection from blood pressure knowledge questionnaire and medication adherence. All this data will be shared via excel data files, and the results from all clinical evaluations will be shared. Excel software and Microsoft word software will be needed to share and view these data files.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 YEARS